CLINICAL TRIAL: NCT06353945
Title: Perceived Effectiveness of the Vaginal Moisturizer Investigational Product Under Normal Conditions of Use.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herbarium Laboratorio Botanico Ltda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HB062-24
Record Dates: First submitted 2024-03-28; First posted 2024-04-09 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Vaginal Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vaginal moisturizer (Experimental): 45 participants treated with vaginal moisturizer
  Interventions: Device: vaginal moisturizer

INTERVENTIONS:
Device: vaginal moisturizer — vaginal moisturizer

SUMMARY:
The present research project aims to evaluate the perceived effectiveness of the product under investigation under normal conditions of use for 28 days, to defend the claims "High hydration power, relief of discomfort and improvement of vaginal tone."

DETAILED DESCRIPTION:
This research project aims to evaluate the perceived efficacy of the product under investigation under normal conditions of use for 28 days, to defend the attributes expected for this product category. The study will be carried out through the application of questionnaires, which will be answered by the participants. The study will be conducted with a Brazilian sample in which 45 research participants will be included.

ELIGIBILITY:
Inclusion Criteria:

1. Age range between 25 and 70 years old.
2. Phototypes: I to IV, according to Fitzpatrick classification;
3. Sex: female
4. Intact skin in the evaluation region.
5. Participants complaining of vaginal dryness;
6. Agree to adhere to the study procedures and requirements: study time, return(s) to the laboratory to perform study procedures, home use of the investigational product, filling out the usage diary, not changing cosmetic habits during the study period .
7. Agree not to carry out dermatological or aesthetic treatments until the end of the study and agree not to use any products from the same category as the investigational product.
8. Signing of the Free and Informed Consent Form (TCLE).

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. Skin marks in the experimental area that interfere with the assessment of possible skin reactions.
3. Active dermatoses (local or disseminated) that could interfere with the study results.
4. History of ineffectiveness, allergic reactions, irritation or intense sensation of discomfort to topical products: health products or medications.
5. Expected vaccination during the study or up to 3 weeks before the study;
6. Not taking vitamin A (acid and/or its derivatives orally or topically up to 1 month before the start of the study.)
7. Patients with immunodeficiencies.
8. History of atopy (atopic dermatitis, allergic rhinitis, allergic bronchitis, allergic conjunctivitis, etc.).
9. Use of non-steroidal anti-inflammatory drugs, corticosteroids, antihistamines, photosensitizers or immunosuppressants up to 2 weeks before the study (or considering depot corticosteroids, the interval should be 1 month before the selection).
10. Aesthetic or dermatological treatment up to 4 weeks before the study.
11. Hormonal treatments not stable in the last 3 months.
12. Hyperpigmentation associated with the use of drugs such as tetracyclines, phenothiazides or amiodarone.
13. Hyperpigmentation associated with photosensitivity.
14. People directly involved in carrying out this study and their families.
15. History of lack of adherence or unwillingness to adhere to the study protocol.
16. Any condition that, in the researcher's opinion, could compromise the study.
17. Be participating in another study in the same region of application.

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
evaluate the perceived effectiveness of the investigational product | 28 days
  The perceived efficacy of the subjective method will be evaluated by means of questionnaires answered by the research participants after the first use and 28 days of use of the investigational product using a rating scale. The results of this evaluation will be used to analyze the frequency of scores for each attribute evaluated. Based on the results of the evaluation of the product's efficacy, an analysis of the frequency of scores for each question evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Kosmoscience Ciência e Tecnologia Cosmética Ltda, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No